CLINICAL TRIAL: NCT00358410
Title: An Exploratory Study to Investigate the Effects of the NK1 Antagonist GW679769, 60 mg Once Daily for 4 Days, on Gastric Accommodation, Gastric Emptying and Gastric Distension-induced Perception and Discomfort in Adult Male and Female Patients With Functional Dyspepsia, in a Single Center, Placebo-controlled, Double-blind, Randomised, Two-period Crossover Study
Brief Title: An Exploratory Study Examining The Effects Of Taking GW679769 Once-Daily For 4 Days In Patients With Functional Dyspepsia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: GW679769/904
Record Dates: First submitted 2006-07-27; First posted 2006-07-31 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Nonulcer Dyspepsia
Keywords: Functional Dyspepsia; Barostat; Stomach
MeSH Terms: interventions — casopitant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GW679769 (Experimental): 120mg once a day
  Interventions: Drug: GW679769 oral tablets
- Placebo (Placebo Comparator): Placebo once a day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW679769 oral tablets — 2x GW679769 60mg tablets
  Arms: GW679769
Drug: Placebo — Placebo oral tablets to match experimental intervention
  Arms: Placebo

SUMMARY:
This study was designed is to examine the idea that GW679769 has an effect on three of the pathophysiological disturbances reported in patients with Functional Dyspepsia (FD): impaired stomach accommodation to a meal, delayed stomach emptying, and visceral hypersensitivity to distension.

DETAILED DESCRIPTION:
An exploratory study to investigate the effects of the NK1 antagonist GW679769, 120 mg once daily for 4 days, on gastric accommodation, gastric emptying and gastric distension-induced perception and discomfort in adult male and female patients with functional dyspepsia, in a single-centre, placebo-controlled, double-blind, randomised, two-period crossover study

ELIGIBILITY:
Inclusion criteria:

* Functional dyspepsia as diagnosed according to the Rome II criteria
* Must had a one month trial (full dose) of proton pump inhibitor treatment within the last 6 months, during a symptomatic period, that produced no lasting response, although this may not be required for those patients who have no symptoms of heartburn and do not present pain-predominant dyspepsia symptoms. Such decision will be left to the Principal Investigator's discretion.
* Patients who are non-smokers or smokers who smoke up to 20 cigarettes per day

Exclusion criteria:

* Active or history of peptic ulcer disorder
* History of major abdominal surgery
* History of underlying psychiatric illness, or current active psychiatric morbidity
* Pregnant or nursing women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
To identify whether GW679769 has an effect on gastric accommodation to a meal, as measured by gastric barostat in male and female patients with FD. Meal induced fundus relaxation as measured by gastric barostat. | Three to Five Days

SECONDARY OUTCOMES:
Rate of gastric emptying as measured by dual breath test.Thresholds for perception and discomfort during gastric distension by gastric barostat. | Three to Five days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Leuven, Belgium